CLINICAL TRIAL: NCT02716558
Title: A Clinical Trial to Assess the Retention and Caries Preventive Effects of Moisture Tolerant Resin Sealant and ART Sealants
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Dr. Praveen B.H (Other)
Collaborators: Nathajirao G. Halgekar Institute of Dental Sciences & Research centre, Karnataka, India (Unknown)
Responsible Party: Sponsor-Investigator, Dr. Praveen B.H, Principal investigator, Kamineni Institute of Dental Sciences
Organization: Kamineni Institute of Dental Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: AIMST university
Record Dates: First submitted 2016-03-07; First posted 2016-03-23 (Estimated); Last update posted 2018-06-26 (Actual); Status verified 2018-06

CONDITIONS: Retention

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Moisture tolerant resin sealant (Experimental): Moisture resistant sealant (wet bond sealant)
  Interventions: Other: Resin sealant application
- ART sealant (Active Comparator): Glass inomer based sealant
  Interventions: Other: ART Sealant Application

INTERVENTIONS:
Other: ART Sealant Application — application of the ART sealant using high viscosity glass inomer cements.
  Arms: ART sealant
Other: Resin sealant application — application of the moisture tolerant sealant according to the manufacturers instructions.
  Arms: Moisture tolerant resin sealant

SUMMARY:
It is a clinical trial which employs a split mouth design to assess the retention of a moisture tolerant resin based sealant and the ART(Atraumatic restorative treatment) sealants on a representative sample of 7- 12 year old school children of a district in Belgaum, Karnataka, India.

DETAILED DESCRIPTION:
Dental caries is a diet dependent, transmissible, micro biologically mediated disease, which follows both an infectious and chronic disease model that progresses slowly with periods of quiescence.

From the literature available, it is understood that although dental caries is on the decline in many of the developed countries, it still remains unchanged with regards to pits and fissure caries of occlusal surfaces of the teeth. This increase in susceptibility is due to its inherent morphological structure which makes a person unable to maintain cleanliness devoid of food lodgement.. Although pits and fissures of occlusal surfaces form only 12.5% of all tooth surfaces yet, they constitute more than 2/3rd of total caries experience among young permanent teeth.

The prevention of dental caries not only includes measures to prevent the occurrence of disease, such as risk factor reduction, but also to arrest the progress of disease and reduce the consequences of disease once it is established Creativity in this effort against fissure caries continues, with newer materials and technology tested each year. The traditional preventive methods, such as diet control and fluoride therapy effectively prevent dental caries on smooth tooth surfaces, but they have not been satisfactory methods to control caries in pit and fissures.

At the time that acid etch bonding was first described by Buonocore in 1955 , bonding was a new technology, and a logical step in its use was the prevention of pit and fissure decay. The focus of Buonocore's work was the development of a sealant to prevent occlusal caries on posterior teeth.Thus, resin sealants were born. Acid treatment of enamel or dentin, whether a priory or concomitant bonding step, has been integrated into methods to retain materials and significantly reduce micro leakage at material tooth interfaces.

Pit and fissure sealant is a "cement or resin material which is introduced into unprepared occlusal pit and fissure of caries susceptible teeth, forming a mechanical and physical protective layer against the action of acid producing bacteria and their substrate".

Pit and fissure sealants introduced by Cueto and Buonocore in 1967 have been accepted as an efficient caries preventive method. For most of the period since the introduction of the sealants, the focus has been on Bis-GMA resin based materials. Resin based sealants have been tested on many occasions and have generally been shown to be an effective method of caries prevention for children and young adults,. The efficacy of these resin sealants in preventing caries has been associated with the duration and degree of sealant retention.

However, the application of resin based sealants demands total moisture control as they are hydrophobic in nature and is often only possible to a limited extent particularly in children with low compliance. Ideally, a material combining the attributes of resin based sealants, such as good retention and good physical properties with moisture tolerance would be desirable.

Recently, a unique moisture tolerant resin based sealant called the embrace wet bond sealant has been introduced. Embrace incorporates di-tri and multi-functional acrylate monomers into an advanced acid integrating chemistry that is activated by moisture. The advantages are wet bonding, tooth integrating, better retention, superior marginal seal, less technique sensitive and increased fluoride release.

Another class of sealants that have been developed are the glass inomer based sealants and these are primarily indicated for subjects, where in total moisture control is not achievable. These sealants, although being hydrophilic have a major drawback which is the low retentivity. In order to overcome this drawback, high viscosity glass inomer cements using the ART approach have been introduced as sealant materials.

A notable point which has been to be given further consideration is the fact that although the embrace wet bond sealant (resin based sealant) and the ART sealant (GIC based sealant) belong to different classes of sealants, they can be indicated in conditions where total moisture control is impossible to achieve.

There is an absolute lack of information regarding the relative performance of the moisture tolerant resin based sealant (embrace wet bond sealant) against the ART sealants and therefore this clinical trial will evaluate the retention and the caries preventive aspect of the above said materials among a representative sample of 7- 10 year old caries prone children.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with fully erupted contralateral permanent mandibular first molars with well defined deep irregular pits and fissures. The entire tooth surface should be visible in the mouth and free of mucosal tissue.

Exclusion Criteria:

* An open carious lesion exists.
* A large occlusal restoration if already present.
* Presence of caries on the other surfaces of the same tooth.
* Subjects with developmental anomalies and hypoplastic permanent first molars.
* Subjects who were suffering from any systemic disease or those who were on any long term medication.

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 93 (Actual)
Dates: Start 2016-02; Primary Completion 2017-03 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Retention of the sealants | Baseline to 1 year
  The retention of the sealants will be assessed by using the MODIFIED SIMENSONS CRITERIA

CONTACTS AND LOCATIONS:
Overall Officials: Praveen Bhoopathi, M.D.S, Study Director — Lecturer
Locations (1):
- Maratha Mandal's Nathajirao G. Halgekar Institute of Dental Sciences & Research Centre., Belagavi, Karnataka, India

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Haricharan PB, Barad N, Patil CR, Voruganti S, Mudrakola DP, Turagam N. Dawn of a New Age Fissure Sealant? A Study Evaluating the Clinical Performance of Embrace WetBond and ART Sealants: Results from a Randomized Controlled Clinical Trial. Eur J Dent. 2019 Oct;13(4):503-509. doi: 10.1055/s-0039-1696894. Epub 2019 Dec 31. PMID 31891967